CLINICAL TRIAL: NCT02770131
Title: Observational Serial Chart Review of Repatha® Use in European Subjects With Hyperlipidaemia
Brief Title: Chart Review of Repatha® in Subjects With Hyperlipidaemia
Acronym: HEYMANS
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130296
Record Dates: First submitted 2016-04-27; First posted 2016-05-12 (Estimated); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Hypercholesterolaemia
Keywords: hypercholesterolaemia; lipid-lowering therapies
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: To describe the clinical characteristics of subjects at initiation of Repatha® (up to 2000 subjects).

SUMMARY:
Review of clinical characteristics of patients who are prescribed Repatha® and how their treatment is managed.

ELIGIBILITY:
Inclusion Criteria:

Adults (>18 years) Provided informed consent Initiated on Repatha® at physician's discretion, after 1st August 2015 Received at least one dose of Repatha®

Exclusion Criteria:

Enrolled in an interventional study of PCSK9 inhibitor within 12 weeks prior to initiation of Repatha® Received commercially available PCSK9 inhibitor within 12 weeks prior to initiation of Repatha®

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients from European countries, who have received Repatha® as part of routine clinical management of their hyperlipidaemia, between August 2015 and June 2021.
Sampling Method: Probability Sample
Enrollment: 1986 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Description of clinical characteristics of subjects initiated on Repatha® | Study day 1
  Age at initiation of Repatha®, Gender Familial hypercholesterolaemia status Diabetic status, Cardiovascular history History of statin intolerance

SECONDARY OUTCOMES:
Describe LDL-C and other cholesterol values over time | Up to 26 weeks prior to the first dose of Repatha®, up to 30 months post first dose of Repatha®
  Detail all cholesterol assessments recorded during the observation period (Total Cholesterol, LDL-C, HDL-C, Non-HDL-C and Triglycerides).
Describe Repatha® dose over time | From the first dose of Repatha® up to 30 months post first dose
  Record Repatha® dose in mg
Describe use of other lipid-modifying therapies | From the first dose of Repatha® up to 30 months post first dose
  Describe lipid-modifying therapies over time, type, dose and dose frequency during the observation period
Describe Physician visits | From the first dose of Repatha® up to 30 months post first dose
  Collection of all primary and secondary healthcare visit dates and classification as to cardiovascular and non-cardiovascular.
Describe hospitalizations | From the first dose of Repatha® up to 30 months post first dose
  Detail all hospitalizations from enrolment to end of study
Describe Repatha® dose frequency over time | From the first dose of Repatha® up to 30 months post first dose
  Record dose frequency (Q2W, QM)
Describe Repatha® administrative device use over time | From the first dose of Repatha® up to 30 months post first dose
  Record Repatha® administration device details, personal injector, autoinjector or pre-filled syringe throughout the observation period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (144):
- Austria (8):
  - Research Site, Feldkirch
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Villach
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, La Louvière
  - Research Site, Leuven
- Bulgaria (6):
  - Research Site, Kostenets
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Czechia (9):
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Hradec Králové
  - Research Site, Liberec
  - Research Site, Olomouc
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Ústí nad Labem
  - Research Site, Zlín
- Germany (32):
  - Research Site, Aachen
  - Research Site, Bad Reichenhall
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bochum
  - Research Site, Borsdorf
  - Research Site, Detmold
  - Research Site, Garbsen
  - Research Site, Germering
  - Research Site, Göttingen
  - Research Site, Halberstadt
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Langenhagen
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Markleeberg
  - Research Site, Mönchengladbach
  - Research Site, Mühldorf
  - Research Site, Mülheim
  - Research Site, München
  - Research Site, Neuwied
  - Research Site, Nuremberg
  - Research Site, Oschatz
  - Research Site, Pirna
  - Research Site, Potsdam
  - Research Site, Rostock
  - Research Site, Rotenburg (Wümme)
  - Research Site, Viersen-Dülken
  - Research Site, Villingen-Schwenningen
  - Research Site, Zwickau
- Greece (7):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Italy (30):
  - Research Site, Acerra
  - Research Site, Arzignano
  - Research Site, Asti
  - Research Site, Bassano Del Grappa (VI)
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Brindisi
  - Research Site, Catanzaro
  - Research Site, Cinisello Balsamo (MI)
  - Research Site, Cona FE
  - Research Site, Cosenza
  - Research Site, Foggia
  - Research Site, Lido Di Camaiore LU
  - Research Site, Messina
  - Research Site, Mestre (VE)
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pescara
  - Research Site, Reggio Calabria
  - Research Site, Rivoli
  - Research Site, Roma
  - Research Site, Salerno
  - Research Site, Seriate
  - Research Site, Sesto San Giovanni (MI)
  - Research Site, Taranto
  - Research Site, Torrette Di Ancona
  - Research Site, Treviglio (BG)
  - Research Site, Trieste
- Portugal (6):
  - Research Site, Almada
  - Research Site, Carnaxide
  - Research Site, Coimbra
  - Research Site, Faro
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
- Slovakia (18):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Handlová
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Martin
  - Research Site, Moldava nad Bodvou
  - Research Site, Myjava
  - Research Site, Námestovo
  - Research Site, Nitra
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Trnava
  - Research Site, Žilina
- Spain (14):
  - Research Site, Cadiz, Andalusia
  - Research Site, Huelva, Andalusia
  - Research Site, Jaén, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Reus, Catalonia
  - Research Site, Sabadell, Catalonia
  - Research Site, Ferrol, Galicia
  - Research Site, Lugo, Galicia
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Madrid
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala
- Switzerland (5):
  - Research Site, Basel
  - Research Site, Geneva
  - Research Site, Lugano
  - Research Site, Winterthur
  - Research Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Ray KK, Dhalwani N, Sibartie M, Bridges I, Ebenbichler C, Perrone-Filardi P, Villa G, Vogt A, Bruckert E. Low-density lipoprotein cholesterol levels exceed the recommended European threshold for PCSK9i initiation: lessons from the HEYMANS study. Eur Heart J Qual Care Clin Outcomes. 2022 Jun 6;8(4):447-460. doi: 10.1093/ehjqcco/qcac009. PMID 35175350
- [Background] Blaha V, Margoczy R, Petrov I, Postadzhiyan A, Raslova K, Rosolova H, Bridges I, Dhalwani NN, Zachlederova M, Ray KK. Evolocumab is Initiated in Central and Eastern Europe at Much Higher LDL-C Levels Than Recommended in Guidelines: Results from the Observational HEYMANS Study. J Cardiovasc Pharmacol Ther. 2023 Jan-Dec;28:10742484231172847. doi: 10.1177/10742484231172847. PMID 37218974
- [Background] Blanco Echevarria A, Garcia Diaz JD, Caixas A, Plana Gil N, Rico Corral MA, Bridges I, Dhalwani N, Gatell Menchen S, Ray KK. Long-term treatment persistence and maintained reduction of LDL-cholesterol levels with evolocumab over 30 months: Results from the Spanish cohort of the European prospective HEYMANS study. Clin Investig Arterioscler. 2023 Nov-Dec;35(6):263-271. doi: 10.1016/j.arteri.2023.04.004. Epub 2023 May 24. English, Spanish. PMID 37236829
- [Background] Ebenbichler C, Drexel H, Hanusch U, Toplak H, Dhalwani NN, Bridges I, Hoelzl R, Hemetsberger M, Ray KK. Evolocumab effectiveness in the real-world setting: Austrian data from the pan-European observational HEYMANS study. Wien Klin Wochenschr. 2024 Feb;136(3-4):77-86. doi: 10.1007/s00508-023-02245-w. Epub 2023 Jul 31. PMID 37525072
- [Background] Sudano I, Krahenbuhl S, Mach F, Anstett A, Dhalwani N, Bridges I, Sibartie M, Ray KK. Evolocumab use in clinical practice in Switzerland: final data of the observational HEYMANS cohort study. Ther Adv Cardiovasc Dis. 2024 Jan-Dec;18:17539447231213288. doi: 10.1177/17539447231213288. PMID 38183273
- [Background] Lehrke M, Vogt A, Schettler V, Girndt M, Fraass U, Tabbert-Zitzler A, Bridges I, Dhalwani NN, Ray KK. Evolocumab-Based LDL-C Management in High and Very High Cardiovascular Risk Patients in German Clinical Practice: The HEYMANS Study. Adv Ther. 2024 Mar;41(3):1184-1200. doi: 10.1007/s12325-023-02757-x. Epub 2024 Jan 30. PMID 38286961
- [Background] Vlachopoulos C, Massia D, Kochiadakis G, Kolovou G, Patsilinakos S, Bridges I, Sibartie M, Dhalwani NN, Liberopoulos E, Ray KK. Evolocumab use in Greece is associated with early and sustainable reductions in low-density cholesterol (LDL-C) and high persistence to therapy: Results from the Greek cohort analysis of the observational HEYMANS study. Hellenic J Cardiol. 2023 Nov-Dec;74:74-76. doi: 10.1016/j.hjc.2023.09.003. Epub 2023 Sep 18. No abstract available. PMID 37730147
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com